CLINICAL TRIAL: NCT02888145
Title: Investigating Minimal Residual Disease in Autopreserved Ovarian Tissue in Cases of Neoplastic Pathology
Acronym: OVAGRAFT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: CHU de Reims (Other); University Hospital, Marseille (Other); University Hospital, Lille (Other); Central Hospital, Nancy, France (Other); University Hospital, Grenoble (Other); CMCO SIHCUS, Schiltingheim (Other); University Hospital, Bordeaux (Other); University Hospital, Limoges (Other); Nantes University Hospital (Other); University Hospital, Toulouse (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: P/2012/154
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2018-01

CONDITIONS: Neoplastic Pathology; Autopreserved Ovarian Tissue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Cryopreservation of ovarian tissue is offered to young girls and women aged under 35 who have to undergo sterilizing gonadotoxic treatment, with the aim of preserving their fertility. The main part of the ovary is preserved, as primordial and primary follicles are resistant to freezing / thawing protocols. In the absence of other techniques (in vivo maturation, injecting isolated ovarian follicles, etc.) autografting this cryopreserved tissue is currently the only technique allowing fertility to be restored. Autograft is possible only if the indication for ovary cryopreservation is a non-neoplastic pathology or a malignant pathology with a low risk of ovarian metastasis. In other cases of neoplastic pathologies, particularly in cases of acute leukemia, tissue cannot as yet be re-used due to the lack of any codified technique for evaluating residual disease (MRD). The team has for two years been developing and validating a technique to look for residual disease in fragments of ovarian cortex in cases of acute leukemia. This technique is based on an original protocol for dissociating ovarian tissue to obtain a population of isolated ovarian cells that may be analyzed by multicolor flow cytometry. The specificity and sensitivity of the technique have been demonstrated in an experimental model. This model consists in using 8 color flow cytometry to look for characterizable leukemia cells added in different dilutions to a population of isolated ovarian cells taken from model ovarian cortex and up to a dilution of 10-5. When the molecular markers were present on diagnosis, they were found by RQ-PCR (Real-Time Quantitative Polymerase Chain Reaction) with the same dilutions. The model tissue came from laparoscopic ovarian drilling in patients with polycystic ovary syndrome. The main objective of this project is to validate techniques that have been previously codified with different populations of leukemia cells that may be characterized. We then aim to adapt and validate this technique to look for MRD using 8 color flow cytometry on cryopreserved fragments of ovarian cortex from leukemia patients that are at risk of metastasis. Secondary objectives will be to implement procedures for oncological qualification of grafts in cases of malignant pathology and to consider the recommendations for using this cryopreserved ovarian tissue through the autograft technique for these indications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have cryopreserved their ovarian tissue
* Patients with premature ovarian insufficiency
* Patients aged from 18 to 43 years for the restoration of ovarian function
* No objection from the patient
* Patients who have already received ovarian tissue autograft

Exclusion Criteria:

* Patients aged Under 18 years (bone age)
* Patients older than 43 years
* Patient refusing to be included
* Patients (adults) Under guardianship, curators and safeguard justice

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients likely to re-use their cryopreserved ovarian tissue by autograft
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Amount of MRD detected using 8 colors flow cytometry on cryopreserved fragments of ovarian cortex from leukemia patients that are at risk of metastasis | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roux C, Amiot C, Agnani G, Aubard Y, Rohrlich PS, Piver P. Live birth after ovarian tissue autograft in a patient with sickle cell disease treated by allogeneic bone marrow transplantation. Fertil Steril. 2010 May 1;93(7):2413.e15-9. doi: 10.1016/j.fertnstert.2009.12.022. Epub 2010 Feb 1. PMID 20117783
- [Background] Amiot C, Angelot-Delettre F, Zver T, Alvergnas-Vieille M, Saas P, Garnache-Ottou F, Roux C. Minimal residual disease detection of leukemic cells in ovarian cortex by eight-color flow cytometry. Hum Reprod. 2013 Aug;28(8):2157-67. doi: 10.1093/humrep/det126. Epub 2013 Apr 30. PMID 23633552
- [Background] Fauque P, Ben Amor A, Joanne C, Agnani G, Bresson JL, Roux C. Use of trypan blue staining to assess the quality of ovarian cryopreservation. Fertil Steril. 2007 May;87(5):1200-7. doi: 10.1016/j.fertnstert.2006.08.115. Epub 2007 Feb 20. PMID 17307173
- [Background] Zver T, Alvergnas-Vieille M, Garnache-Ottou F, Roux C, Amiot C. A new method for evaluating the risk of transferring leukemic cells with transplanted cryopreserved ovarian tissue. J Assist Reprod Genet. 2015 Aug;32(8):1263-6. doi: 10.1007/s10815-015-0512-4. Epub 2015 Jul 3. PMID 26139154
- [Background] Zver T, Alvergnas-Vieille M, Garnache-Ottou F, Ferrand C, Roux C, Amiot C. Minimal residual disease detection in cryopreserved ovarian tissue by multicolor flow cytometry in acute myeloid leukemia. Haematologica. 2014 Dec;99(12):e249-52. doi: 10.3324/haematol.2014.113373. Epub 2014 Sep 19. No abstract available. PMID 25239266